CLINICAL TRIAL: NCT02602067
Title: A Dose Escalation Study to Evaluate Safety, Tolerability Dosimetry, Pharmacokinetics and Preliminary Efficacy of 131I-Tenatumomab Treatment in Tenascin-C Positive Cancer Patients
Brief Title: 131Iodine-Tenatumomab Treatment in Tenascin-C Positive Cancer Patients
Acronym: Tenatumomab
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Uptake of drug into the tumour lesion was negligible
Sponsor: sigma-tau i.f.r. S.p.A. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TENATUMOMAB/ST2146-CR-14-001; 2014-003832-38 (EudraCT Number)
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-01

CONDITIONS: Breast Neoplasm; Head and Neck Neoplasm; Skin Neoplasm; Respiratory Tract Neoplasm; Urogenital Neoplasm; Digestive System Neoplasm; Pancreatic Neoplasm; Connective and Soft Tissue Neoplasm; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Skin Neoplasms; Respiratory Tract Neoplasms; Urogenital Neoplasms; Digestive System Neoplasms; Pancreatic Neoplasms; Neoplasms, Connective and Soft Tissue; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: Tenatumomab infusion
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 131I-Tenatumomab (Experimental): Diagnostic: each patient will receive one single i.v. infusion of 370 MBq±10% 131I-Tenatumomab in 10 ml of saline (conveyed by 10 ±10%, 20 ±10%, 40 ±10% mg of Tenatumomab). It will be administered as a short infusion in approximately 30 minutes (333 ° µl / min).
  Therapeutic: each patient will receive one single i.v. infusion, escalating 131I-Tenatumomab dose starting at 2.5 GBq±10%,with escalation steps of 1 GBq, up to 5.5 GBq±10% in 10 ml of saline, (conveyed by 10 ±10% , 20 ±10%, 40 ±10% mg of Tenatumomab). It will be administered as a short infusion in approximately 30 minutes (333° µl / min)
  Interventions: Combination Product: 131I-Tenatumomab

INTERVENTIONS:
Combination Product: 131I-Tenatumomab — I131anti-Tenascin monoclonal antibody administered to be targeted on neoplasms expressing Tenascin-C
  Other Names: Tenatumomab/ST2146

SUMMARY:
Tenatumomab is a Sigma-Tau developed new anti-Tenascin antibody. It is a murine monoclonal antibody directed towards Tenascin-C. By means of this antibody, Tenascin-C expression was studied on a commercial tissue array slides each carrying malignant breast, colorectal, lung, ovarian or B and T cell Non-Hodgkin Limphoma tissue sections. All these cancers type showed positivity to Tenascin-C between the 64% and 13.3%. Consequently, Sigma-tau is exploring the use of the 131I-labeled Tenatumomab for anti-cancer radioimmunotherapy.

DETAILED DESCRIPTION:
This will be an open-label dose escalation study. The study will be conducted in two steps:

1. STEP A aims to identify the optimal amount of antibody to convey the specific radio-label activity of radionuclide.
2. STEP B will be conducted with the amount of antibody chosen in STEP A, and an escalating radio-labeled therapeutic dose response curve will be performed (3.5 to 5.5 GBq) A maximum of 36 evaluable patients suffering from treatment-refractory Tenascin-C positive tumors.

This dose escalation study will be evaluated using descriptive statistics: no sample size calculation was performed

Primary objectives

1. To identify the Maximum Tolerated Dose (MTD) and assess Safety and Tolerability of i.v. infused 131I-Tenatumomab.
2. To identify the optimal amount of unlabeled Tenatumomab able to convey 131I- Tenatumomab with the highest Tumor/nonTumor ratio.
3. To evaluate the whole body Dosimetry (safety dosimetry) and Tumor to normal tissue ratio (T/nT ratio, referred to AUC) of i.v.infused 131I-Tenatumomab.
4. To evaluate intra-lesional distribution and retention of 131I-Tenatumomab and to record individual lesion dosimetry.
5. To evaluate systemic biodistribution, pharmacokinetics, urinary excretion and dose linearity of 131I-Tenatumomab.

Secondary objectives

1. To evaluate proportional 131I-Tenatumomab tumor binding, as a function of the total load.
2. To evaluate Pharmacokinetics of Tenatumomab (protein and protein related materials) in serum.
3. To evaluate preliminary Efficacy of 131I-Tenatumomab based on disease response rate (Complete Response, Partial Response, Stable Disease) and patient's general clinical condition by ECOG performance status assessment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent.
* 2. A patient who has (a) a histologically documented advanced tumor that has relapsed from, or is refractory to, standard treatment and for which no other standard treatment is available and (b) confirmed Tenascin-C expression obtained through a biopsy on at least one reachable tumor lesion.

These patients will have failed one or more prior therapeutic line and had assessable and measurable disease expression, but were not considered eligible for other standard approaches with curative intent, as assessed by the Investigator.

* 3. Agreement to hemopoietic stem cell collection procedures (the procedure will be performed upon clinical evaluation of the Investigator and if deemed necessary in the interest of the patient).
* 4. Male or female ≥18 years of age
* 5. Eastern Cooperative Oncology Group (ECOG), or WHO performance status of ≤ 2 or Karnofsky > 60
* 6. Life expectancy of at least 3 months.
* 7. Negative pregnancy test for all women of child-bearing potential. Appropriate contraception (one highly effective method or a combination of acceptable methods) is to be used during the study period and until 90 days after the last follow-up visit (End of Study Visit)
* 8. Hematological, thyroid, liver, cardiac and renal function test results ≤ grade 2 toxicity (according to US National Cancer Institute's "Common Terminology Criteria for Adverse Events v4.03 [CTCAE]"), e.g.:

Haematology:

* Hematocrit ≥ 30%
* Hemoglobin ≥ 9.0 g/dl
* White blood cell count ≥ 3 x 109/L
* Neutrophils > 1.5 x109/L
* Platelets ≥ 100x 109/L

Thyroid:

- Free-Triiodothyronine and Free-Thyroxine ≤ 3 times upper limit of normal or >3 times lower limit of normal.

Liver:

* Alanine transaminase, Aspartate transaminase, Alkaline Phosphatase ≤ 2.5 times institutional upper limit of normal (ULN) or ≤5 x ULN in presence of liver metastases.
* Bilirubin ≤ 1.5 x ULN or ≤3 x ULN in presence of liver metastases.

Renal:

* Urine protein: ≤30 mg/dl or dipstick: ≤3
* eGFR≥60 ml/min/1.73 m2 (with Chronic kideny disease-Epidemiology collaboration formula)

Cardiac

• Resting Ejection Fraction (EF) ≥ 50%

Exclusion Criteria:

* 1. Known hypersensitivity to Tenatumomab, Iodine or any excipient.
* 2. Active infection at screening or history of severe infection within the previous 2 months, if considered clinically relevant by the Investigator.
* 3. Positive test to Human Immunodeficiency Virus (HIV) and/or chronically active Hepatitis B or C.
* 4. Patients with primary Central nervous system tumor or cerebral metastases.
* 5. Administration of another investigational medicinal product within 45days before the screening period.
* 6. Previous treatment with any radiopharmaceutical within a period corresponding to 8 half-lives of the radionuclide used prior to the administration of study drug.
* 7. History of somatic or psychiatric disease/condition that may interfere with the objectives of the study.
* 8. Major illness, trauma, or surgery within 2 weeks before the screening period, if considered clinically significant by the Investigator.
* 9. Patient who underwent chemotherapy and/or radiation therapy and/or treatments with biologics (which are not to be of murine origin) within 4 weeks before the screening period.
* 10. Women who are breast feeding, due to the potential risk of damage to the infant.
* 11. Men unwilling to use appropriate contraceptive methods during the study and up to 90 days after the last follow-up visit (End of Study Visit).
* 12. Bladder catheterization cannot be performed, or the patient is unwilling to be catheterized if necessary.
* 13. Murine antibodies treated patients. It is at the discretion of the Investigator to exclude patients who have worsened considerably from screening to Day -1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-11; Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity evaluated using NCI Common Toxicity Criteria (CTCAE 4.03) | up to six weeks
  no more details necessary

SECONDARY OUTCOMES:
Adverse Events | up to 1 year
  no more details necessary

OTHER OUTCOMES:
Tumor response | 1 year
  Tumor response according to Response Evaluation Criteria in Solid Tumors RECIST V 1.1 or PERCIST

CONTACTS AND LOCATIONS:
Overall Officials: SECONDO LASTORIA, M.D., Study Chair — ISTITUTO NAZIONALE DEI TUMORI IRCCS - FONDAZIONE "G. PASCALE" NAPLES - ITALY
Locations (7):
- France (3):
  - Institut Bergonnie, Bordeaux
  - Centre Leon Berard, Lyon
  - Icm Val D'Aurelle, Montpellier
- Italy (4):
  - Istituto Nazionale Dei Tumori Irccs - Fondazione "G. Pascale", Naples
  - University of Study of Pisa, Pisa
  - S. Maria Nuova Hospital - Irccs, Reggio Emilia
  - Humanitas Clinical Institute, Rozzano MI